CLINICAL TRIAL: NCT03401801
Title: Impact of Local Anesthetic Volume on Temperature Increase in the Upper Extremity During Ultrasound-guided Stellate Ganglion Block: A Prospective Randomized and Comparative Clinical Trial
Brief Title: Impact of Local Anesthetic Volume During Ultrasound-guided Stellate Ganglion Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Clinical Associate Professor, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1705-101-856
Record Dates: First submitted 2018-01-04; First posted 2018-01-17 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4 ml of 1% lidocaine (Active Comparator): Procedure: 4 ml of 1% lidocaine is injected for stellate ganglion block using the Ultrasound(US)-guided lateral approach at the sixth cervical vertebral level.
  Interventions: Procedure: Stellate ganglion block
- 6 ml of 1% lidocaine (Active Comparator): Procedure: 6 ml of 1% lidocaine is injected for stellate ganglion block using the US-guided lateral approach at the sixth cervical vertebral level.
  Interventions: Procedure: Stellate ganglion block
- 8 ml of 1% lidocaine (Active Comparator): Procedure: 8 ml of 1% lidocaine is injected for stellate ganglion block using the US-guided lateral approach at the sixth cervical vertebral level.
  Interventions: Procedure: Stellate ganglion block

INTERVENTIONS:
Procedure: Stellate ganglion block — Well trained pain physician performs all the ultrasound(US)-guided stellate ganglion block(SGB)s, who is not involved in evaluating study variables. Electrocardiography, noninvasive blood pressure, heart rate, and peripheral oxygen saturation were monitored for all patients before, while, and after conducting procedure. For US-guided SGB, patients are supine positioned, and skin preparation on injection site is done with chlorohexidine. Procedure is conducted under ultrasound guidance at C6 level. 4 ml, 6 ml, and 8 ml of 1% lidocaine is injected for the each group, respectively.

SUMMARY:
The purpose of this study was to compare the temperature changes of the upper extremities when using local anesthetic of various volume (4ml, 6ml, 8ml) in the ultrasound guided stellate ganglion block.

DETAILED DESCRIPTION:
One pain physician performs all US-guided stellate ganglion block(SGB)s, who is not involved in evaluating study variables. Electrocardiography, noninvasive blood pressure, heart rate, and peripheral oxygen saturation were monitored for all patients before, while, and after conducting procedure.

For US-guided SGB, patients are supine positioned, and skin preparation on injection site is done with chlorohexidine. Procedure is conducted under ultrasound guidance at C6 level. 4ml, 6ml, and 8ml of 1% lidocaine is injected for the each group, respectively. Syringes are prepared by one nurse who do not involved in other steps of this study.

Temperature measurement is conducted 4 times (before US-guided SGB and after 10, 20, and 30m from SGB) at both hands, face, axillar by one person who's not involved in other measuring in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 85 years
* Patients with a new or known diagnosis of chronic neuropathic pain at the upper extremity or face.

Exclusion Criteria:

* Refusal of a patient
* Any vascular disease in the upper extremities (or face)
* Previous history of thoracic sympathetic or stellate ganglion neurolysis (e.g. thermocoagulation, radiofrequency neuromodulation, and/or chemical neurolysis)
* Coagulopathy
* Systemic infection or local infection at the needle injection site
* Major deformation at the level of the neck (radiotherapy, surgery, etc.)
* Concomitant chronic pain syndrome at other sites.
* Post-pneumonectomy on the controlateral side
* Known allergy to local anesthetics of amide type
* Inability to understand a numeric rating pain scale (cognitive dysfunction)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-07-21 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Temperature change(°C) in ipsilateral arm | thirty minute after US-guided SGB
  Temperature is measured with a laser thermometer on the palmar aspect of 3 cm below from the middle finger.

SECONDARY OUTCOMES:
Temperature changes(°C) in ipsilateral arm | 10 and 20 min after US-guided SGB
  Temperature is measured with a laser thermometer on the palmar aspect of 3 cm below from the middle finger.
Temperature changes in ipsilateral face | 10, 20, and 30 min after US-guided SGB
  Temperature is measured with a laser thermometer on a junction between the extended lines from pupil and nostril.
Temperature changes in contralateral face | 10, 20, and 30 min after US-guided SGB
  Temperature is measured with a laser thermometer on a junction between the extended lines from pupil and nostril.
Temperature changes in ipsilateral medial elbow | 10, 20, and 30 min after US-guided SGB
  Temperature is measured with a laser thermometer on the forearm area (3 cm above the medial epicondyle).
Temperature changes in contralateral medial elbow | 10, 20, and 30 min after US-guided SGB
  Temperature is measured with a laser thermometer on the forearm area (3 cm above the medial epicondyle).
Severity of pain using an 11-pointed numerical rating scale(NRS) pain score | Time before block and time of block to 30 minutes after the block
  The pain NRS is a single 11-point numeric scale. An 11-point numeric scale (NRS 11) with 0 representing one pain extreme (e.g., "no pain") and 10 representing the other pain extreme (e.g., "pain as bad as you can imagine" and "worst pain imaginable"). The NRS will be administered verbally or graphically for self-completion. The respondent is asked to indicate the numeric value on the segmented scale that best describes their pain intensity. The number that the respondent indicates on the scale to rate their pain intensity is recorded. Scores range from 0-10. Higher scores indicate greater pain intensity.
Proportion of patients reaching >1.5°C rise of temperature in the ipsilateral arm compared to the contralateral arm | 30 minutes after the block
  Temperature is measured with a laser thermometer on the palmar aspect of 3 cm below from the middle finger.
Proportion of patients reaching >1.5°C rise of temperature in the ipsilateral face compared to the contralateral face | 30 minutes after the block
  Temperature is measured with a laser thermometer on a junction between the extended lines from pupil and nostril.
Proportion of patients with ptosis | 30 minutes after the block
  Check the distance between upper lid margin and light reflex(MRD).

CONTACTS AND LOCATIONS:
Overall Officials: Jee Youn Moon, MD, PhD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kapral S, Krafft P, Gosch M, Fleischmann D, Weinstabl C. Ultrasound imaging for stellate ganglion block: direct visualization of puncture site and local anesthetic spread. A pilot study. Reg Anesth. 1995 Jul-Aug;20(4):323-8. PMID 7577781
- [Background] Schurmann M, Gradl G, Wizgal I, Tutic M, Moser C, Azad S, Beyer A. Clinical and physiologic evaluation of stellate ganglion blockade for complex regional pain syndrome type I. Clin J Pain. 2001 Mar;17(1):94-100. doi: 10.1097/00002508-200103000-00012. PMID 11289093
- [Result] Jung G, Kim BS, Shin KB, Park KB, Kim SY, Song SO. The optimal volume of 0.2% ropivacaine required for an ultrasound-guided stellate ganglion block. Korean J Anesthesiol. 2011 Mar;60(3):179-84. doi: 10.4097/kjae.2011.60.3.179. Epub 2011 Mar 30. PMID 21490819
- [Result] Stevens RA, Stotz A, Kao TC, Powar M, Burgess S, Kleinman B. The relative increase in skin temperature after stellate ganglion block is predictive of a complete sympathectomy of the hand. Reg Anesth Pain Med. 1998 May-Jun;23(3):266-70. doi: 10.1016/s1098-7339(98)90053-0. PMID 9613538